CLINICAL TRIAL: NCT04999891
Title: The Southeast and East Asian Post-Operative Delirium (SEAPOD) Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Sponsor
Other Study IDs: 2020/01350
Record Dates: First submitted 2021-06-24; First posted 2021-08-11 (Actual); Last update posted 2022-10-06 (Actual); Status verified 2022-08

CONDITIONS: Postoperative Delirium; Hip Fractures
Keywords: Geriatrics
MeSH Terms: conditions — Emergence Delirium; Hip Fractures | interventions — Mental Status and Dementia Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Surgical Cohort: Elderly patients aged 65 and above who are planned for hip fracture surgery.
  Interventions: Other: Neurocognitive tests

INTERVENTIONS:
Other: Neurocognitive tests — Battery of neurocognitive tests and questionnaires including MoCA, PHQ-9, Falls History, FIFE, STOPBANG, Nutritional Survey, Global Physical Activity Questionnaire, Brief Pain Index, NuDESC, 3D-CAM.

SUMMARY:
The specific aim of the study will be to investigate the incidences and risk factors for postoperative delirium (POD) after hip fracture surgery in elderly patients aged ≥ 65 years in five different Southeast and East Asian countries.

The secondary objectives are outlined below:

1. To investigate factors in the hospital environments, such as noise levels, ambient lighting, nursing ratios, ward bedding and climate control, that contribute to similarities and/or differences in POD occurrences in different countries and health systems
2. To investigate patient factors, such as disease burden, mental health, education levels, and socioeconomic factors, that contribute to similarities and/or differences in POD occurrences in different countries and health systems
3. To quantify the direct and indirect costs, as well as resource utilization, resulting from the development of POD in each country

DETAILED DESCRIPTION:
Hip fractures encompass all fractures of the upper (proximal) part of the thigh bone (femur). They are commonly divided into two types: intracapsular fractures, which represent those that occur within or proximal to the attachment of the hip joint capsule to the femur, and extracapsular, which represent fractures occurring below or distal to the attachment of the hip joint capsule.

Hip fractures are common in elderly people with an annual incidence rate estimated as 1.29/1000 person-years in men and 2.24/1000 person-years in women. It is the most common condition requiring physical rehabilitation in older adults. The majority (>95%) of people undergo hip surgery following hip fracture. The location of the fracture, stability, and degree of comminution (number of pieces the bone breaks into) determine which operative procedure should be used to repair the hip fracture. The aim of surgery, irrespective of the type of operation, is to reduce pain, facilitate early weight-bearing mobility to improve outcome, and facilitate independence in activities of daily living, such as bathing, dressing, and continence. However, hip fracture is associated with significant pain and loss of independence and function. Although 33-37% of patients return to their prior level of function within six months including those needing assistance, only 24% of people are independently mobile six months after hip fracture.

A major complication in elderly hip fracture patients is POD, with an incidence rate varying from 13% to 65%. POD after hip surgery was significantly associated with non-home discharge disposition, and higher odds of 30-day readmissions and 30-day mortality. POD is also associated with poor outcomes, such as lower rates of immediate postoperative weight bearing, increased pressure sores, and poorer recovery of activities of daily living. In addition, a recent meta-analysis showed that POD after hip surgery translates into long-term cognitive disease burden, by increasing the risk of incident dementia and cognitive decline by a marked odds ratio of 8.957.

No strong evidence exists regarding the treatment of delirium. Several studies performed on delirium prevention in hip fracture patients have described the use of care bundles such as orthogeriatric care and comprehensive geriatric care as an effective potential treatment for this patient group, although the evidence remains weak. However, Inouye et al stated that in the general geriatric population, 30% to 40% of the delirium episodes could be prevented by addressing modifiable risk factors.

Previous studies in the five Asian countries involved in this study show that the incidence of POD after hip fracture surgery varied greatly between countries and within countries: 12.8-27.9% in Japan, 5.07-51.3% in Korea, 13.4-45% in Thailand and 7.2% in Singapore. The incidence of POD in Malaysia can be estimated at 9-12% as reported in the recent HIP Attack trial. However, these studies were heterogenous in terms of patient selection, study methodology and hospital systems. These variations make it difficult to draw a direct comparison regarding the incidence of POD amongst Asian countries and to Western cohorts. Furthermore, the cost of POD to patients and institutions, both direct and indirect, is very poorly defined in Asian countries.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide informed consent
* Elderly patients aged 65 years and above
* Scheduled to undergo elective or emergency hip fracture surgery

Exclusion Criteria:

* History of psychiatric disease
* Baseline cognitive impairment or dementia (MOCA score < 24)
* Illiterate (unable to read or write with local language)
* Active history of substance abuse
* Has a second surgery planned within 5 days of index surgery
* Non-resident of Singapore
* Significant hearing and/or speech impairment
* Planned for admission into the intensive care unit after surgery

Ages: 65 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Elderly patients aged 65 and above scheduled to undergo hip fracture surgery
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2021-08-22 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Development of POD in elderly patients undergoing hip fracture surgery | Before surgery through to 1 year post surgery
  Collection of patient's demographics, medical records and surgical records to establish risk factors for POD development

SECONDARY OUTCOMES:
Healthcare cost of POD in different countries and health systems | Before surgery through to study completion, an average of 1 year
  Quantify the direct and indirect costs, as well as resource utilization, resulting from the development of POD in each country by collecting hospitalization costs
Similarities and/or differences in POD occurrences in different countries and health systems | Before surgery through to 1 year post surgery
  Collection of data such as noise levels, ambient lighting, nursing ratios, ward bedding and climate control, disease burden, mental health, education levels, and socioeconomic factors to establish similarities and/or differences in POD occurrences in different countries and health systems

CONTACTS AND LOCATIONS:
Overall Officials: Lian Kah Ti, Principal Investigator — National University Health System
Locations (13):
- Japan (2):
  - Tohoku University School of Medicine, Sendai
  - Tokyo Women's Medical University, Tokyo
- Malaysia (2):
  - University of Malaya, Kuala Lumpur
  - Universiti Sains Malaysia, Malacca
- Singapore (5):
  - Singapore General Hospital, Singapore
  - Khoo Teck Puat Hospital, Singapore
  - National University Health System, Singapore
  - Ng Teng Fong General Hospital, Singapore
  - Tan Tock Seng Hospital, Singapore
- South Korea (2):
  - Severance Hospital, Seoul
  - St Mary's Hospital, Seoul
- Thailand (2):
  - Ramathibodi Hospital, Bangkok
  - Siriraj Hospital, Bangkok

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Adams AL, Shi J, Takayanagi M, Dell RM, Funahashi TT, Jacobsen SJ. Ten-year hip fracture incidence rate trends in a large California population, 1997-2006. Osteoporos Int. 2013 Jan;24(1):373-6. doi: 10.1007/s00198-012-1938-5. Epub 2012 Feb 21. PMID 22349963
- [Background] Lenze EJ, Skidmore ER, Dew MA, Butters MA, Rogers JC, Begley A, Reynolds CF 3rd, Munin MC. Does depression, apathy or cognitive impairment reduce the benefit of inpatient rehabilitation facilities for elderly hip fracture patients? Gen Hosp Psychiatry. 2007 Mar-Apr;29(2):141-6. doi: 10.1016/j.genhosppsych.2007.01.001. PMID 17336663
- [Background] Uzoigwe CE, Burnand HG, Cheesman CL, Aghedo DO, Faizi M, Middleton RG. Early and ultra-early surgery in hip fracture patients improves survival. Injury. 2013 Jun;44(6):726-9. doi: 10.1016/j.injury.2012.08.025. Epub 2012 Sep 23. PMID 23010072
- [Background] Handoll HH, Cameron ID, Mak JC, Finnegan TP. Multidisciplinary rehabilitation for older people with hip fractures. Cochrane Database Syst Rev. 2009 Oct 7;(4):CD007125. doi: 10.1002/14651858.CD007125.pub2. PMID 19821396
- [Background] Morrison RS, Ahronheim JC, Morrison GR, Darling E, Baskin SA, Morris J, Choi C, Meier DE. Pain and discomfort associated with common hospital procedures and experiences. J Pain Symptom Manage. 1998 Feb;15(2):91-101. PMID 9494307